CLINICAL TRIAL: NCT02537795
Title: Psychiatric Neurosurgery (PNS) for Obsessive Compulsive Disorder (OCD): A Qualitative Analysis of Patient and Family Member Experiences
Status: Recruiting | Type: Observational
Sponsor: Universitaire Ziekenhuizen KU Leuven (Other)
Responsible Party: Sponsor
Other Study IDs: s58187
Record Dates: First submitted 2015-08-21; First posted 2015-09-02 (Estimated); Last update posted 2024-07-10 (Actual); Status verified 2024-07

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Deep Brain Stimulation; Anterior Capsulotomy
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Deep Brain Stimulation

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Deep Brain Stimulation Patients: Patients who have previously been treated with a deep brain stimulation procedure for obsessive compulsive disorder will be included in this group
  Interventions: Device: deep brain stimulation
- Deep Brain Stimulation Family Members: Family members of patients who have previously been treated with a deep brain stimulation procedure for obsessive compulsive disorder will be included in this group
- Anterior Capsulotomy Patients: Patients who have previously been treated with an anterior capsulotomy procedure for obsessive compulsive disorder will be included in this group
  Interventions: Procedure: anterior capsulotomy
- Anterior Capsulotomy Family Members: Family members of patients who have previously been treated with an anterior capsulotomy procedure for obsessive compulsive disorder will be included in this group

INTERVENTIONS:
Device: deep brain stimulation — Electrical stimulation of the anterior limb of the internal capsule or bed nucleus of the stria terminalis
  Groups: Deep Brain Stimulation Patients
Procedure: anterior capsulotomy
  Groups: Anterior Capsulotomy Patients

SUMMARY:
In this study the investigators will use semi-structured interviews to qualitatively analyse patient and family member experiences with either deep brain stimulation or other forms of psychiatric neurosurgery.

ELIGIBILITY:
Inclusion Criteria:

* (family member of) patient who has previously been treated with deep brain stimulation or anterior capsulotomy

Exclusion Criteria:

* none

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: In the University Hospital of Leuven, more than thirty patients suffering from severe OCD have been treated with DBS. The investigators will ask patients who are currently being treated with DBS whether they are willing to participate in this study. The investigators will also ask whether one of their family members might participate, preferentially their partner or another close family member. The aim is to include at least ten patients and their family members. OCD patients, who have been treated with anterior capsulotomy, and their family members will also be asked for participation in this study. The aim is to also include ten patients and family members in this group.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2015-08; Primary Completion 2025-04 (Estimated); Study Completion 2025-04 (Estimated)

PRIMARY OUTCOMES:
Semi-structured Interview | up to 180 months after surgery
  A semi-structured interview of patients and one of their family members will be conducted. Patients and family members will be interviewed separately. The interview will consist of several open ended questions around several themes. The interviews for patients and family members will have their own focus. Patient interviews will focus on living with OCD, living with PNS and the decision making process leading to the PNS procedure. Family member interviews will focus on their own experience in their interaction with OCD patients both before and after PNS

CONTACTS AND LOCATIONS:
Overall Officials: Chris Bervoets, MD, PhD, Principal Investigator — UPC KU Leuven
Locations (1):
- UZ Leuven, Leuven, Vlaams-Brabant, Belgium